CLINICAL TRIAL: NCT01219660
Title: Obstructive Sleep Apnea (OSA) Anesthesia and Positive Airway Pressure
Acronym: OSA
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 091703
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep; apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine if autotitrating positive airway pressure (APAP) naïve patients with OSA can successfully use APAP following general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Obstructive Sleep Apna

Exclusion Criteria:

* non conformers

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)